CLINICAL TRIAL: NCT04174703
Title: Preparing for Eating Disorders Treatment Through Compassionate Letter-Writing
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Allison Kelly, Associate Professor, University of Waterloo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 41135
Record Dates: First submitted 2019-11-04; First posted 2019-11-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Compassion
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder

STUDY DESIGN:
Intervention Model Description: Half of the study participants (n=80) will be placed into the self-compassionate letter-writing intervention group, and half of the study participants (n=80) will be placed into a control group.
Who Masked: Care Provider
Masking Description: The care providers will not be told which condition each participant was assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-compassionate letter-writing intervention (Experimental): An online self-compassionate letter-writing task once per day (10-20 minutes each) for 2 weeks
  Interventions: Other: Self-compassionate letter-writing intervention
- Control condition (No Intervention)

INTERVENTIONS:
Other: Self-compassionate letter-writing intervention — Participants in this condition will be asked to engage in an online self-compassionate letter-writing task once per day (10-20 minutes each) for 2 weeks.
  Arms: Self-compassionate letter-writing intervention

SUMMARY:
Compassion-focused therapy (CFT) seeks to lower shame and help people develop compassion for personal distress and shortcomings. There is increasing evidence to support the benefits of incorporating CFT-based interventions into the treatment of eating disorders (EDs). Building on the investigators' prior research, this study will examine the effects of a two-week CFT-based self-compassion letter-writing intervention on patients with eating disorders. Participants will be recruited from the wait-list of patients scheduled to begin treatment at the outpatient St. Joseph's Healthcare Hamilton Eating Disorders Program, and will be randomly assigned to the two-week letter-writing intervention or to a control group. Results will inform the integration of new empirically-derived interventions into ED treatments to improve the currently dismal rates of ED recovery.

DETAILED DESCRIPTION:
The study consists of two phases. In phase one, participants will be randomly assigned to a two-week daily letter-writing intervention condition or a two-week control condition; phase one will occur two to four weeks prior to the start date of group ED treatment. Participants will complete a brief set of online questionnaires pre-, mid-, and post- two-week condition (i.e. baseline, after one week, and after two weeks).

Following these two weeks of intervention/control condition, all participants will complete a 25-week group treatment program as scheduled by the Eating Disorders Program. For phase two of the study, participants will be asked to complete questionnaires after 5 weeks, after 11 weeks, and post-group treatment. Data that is routinely collected as part of patients' clinical care pre- and post-treatment (i.e. on the first day and last week of group treatment) will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 diagnosis of anorexia nervosa, bulimia nervosa, or binge eating disorder
2. Eligible to start group eating disorders treatment at St. Joseph's Eating Disorder Program
3. 17 years of age or older

Exclusion Criteria: None

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Weight- and Body-Related Shame and Guilt Scale (WEB-SG) | Change from baseline to post-2 weeks of intervention/control condition
  Self-report questionnaire with 12 questions on a 5-point Likert scale (scored 0-4). Total scores range from 0-48, with higher decrease in score indicative of a better outcome (i.e. higher decrease in levels of shame and guilt).
Self-compassion Scale (short form; SCS-SF) | Change from baseline to post-2 weeks of intervention/control condition
  Self-report questionnaire with 12 questions on a 5-point Likert scale (scored 1-5). Total scores range from 12-60, with higher increase in score indicative of a better outcome (i.e. higher increase in levels of self-compassion).
Readiness to Change Eating Behaviours | Change from baseline to post-2 weeks of intervention/control condition
  Self-report questionnaire with 3 questions on a 10-point Likert scale (scored 1-10). Total scores range from 3-30, with higher increase in score indicative of a better outcome (i.e. higher increase in readiness to change disordered eating behaviours).

SECONDARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q) | Change from day 1 to week 25 of group eating disorder treatment
  Self-report questionnaire with 28 questions, collecting two types of data. The EDE-Q collects frequency data of eating disorder behaviours. The EDE-Q also has four subscales assessing the severity of four aspects of ED psychopathology. These subscales are scored using 7-point Likert scales (scored 0-6). Higher decreases in scores are indicative of a better outcome (i.e. higher decreases in eating disorder symptomatology).
Clinical Impairment Assessment (CIA) | Change from day 1 to week 25 of group eating disorder treatment
  Self-report questionnaire with 16 questions on a 4-point Likert scale (scored 0-3). Total scores range from 0-48, with higher decrease in score indicative of a better outcome (i.e. higher decrease in clinical impairment).

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kelly, PhD, Principal Investigator — University of Waterloo
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelly AC, Waring SV. A feasibility study of a 2-week self-compassionate letter-writing intervention for nontreatment seeking individuals with typical and atypical anorexia nervosa. Int J Eat Disord. 2018 Aug;51(8):1005-1009. doi: 10.1002/eat.22930. Epub 2018 Aug 13. PMID 30102787
- [Background] Kelly AC, Wisniewski L, Martin-Wagar C, Hoffman E. Group-Based Compassion-Focused Therapy as an Adjunct to Outpatient Treatment for Eating Disorders: A Pilot Randomized Controlled Trial. Clin Psychol Psychother. 2017 Mar;24(2):475-487. doi: 10.1002/cpp.2018. Epub 2016 May 30. PMID 27237928
- [Background] Kelly AC, Carter JC, Zuroff DC, Borairi S. Self-compassion and fear of self-compassion interact to predict response to eating disorders treatment: a preliminary investigation. Psychother Res. 2013;23(3):252-64. doi: 10.1080/10503307.2012.717310. Epub 2012 Aug 24. PMID 22917037